CLINICAL TRIAL: NCT05503810
Title: Feasibility Randomized Trial of a Social Support Intervention Plus Usual Care Versus Usual Care, Targeting Patients Treated for Cardiac Disease Who Experience Loneliness
Brief Title: Social Support Intervention Targeting Patients Treated for Cardiac Disease Who Experience Loneliness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not feasible. Acceptance rate was too low.
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HeartBuddyPilot
Record Dates: First submitted 2022-08-10; First posted 2022-08-17 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Feasibility
Keywords: Loneliness; Social support; cardiac

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial design with 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Six month social support intervention following in hospital cardiac treatment
  Interventions: Behavioral: Social support
- Control (No Intervention): Regular follow-up

INTERVENTIONS:
Behavioral: Social support — Contact ones a week with Informal caregiver or peer support
  Other Names: Loneliness reduction
  Arms: Intervention

SUMMARY:
Introduction: In patients treated for cardiac disease, loneliness is known to contribute negatively to health behavior, health outcome and increase risk of cardiac and all-cause mortality. Even so, in health care research, social support interventional studies targeting patients who experience loneliness is lacking.

Aim: To determine the feasibility of an individually structured social support intervention targeting patients treated for cardiac disease who experience loneliness.

Design: A feasibility study based on randomized clinical trial design with 1:1 randomization to a 6-month social support program, plus usual care (intervention) versus usual care, (i.e., regular guidelines-based follow-up). Intervention: Patients classified as high risk lonely according to the High Risk Loneliness tool will be provided with an informal caregiver in the six months rehabilitation phase following cardiac disease treatment. The informal caregiver will be designated by the patient from the existing social network or a peer, depending on patients' preferences. The core content of the intervention is through nurse consultations at baseline, one, three and six months, to enhance and reinforce the informal caregiver's competences to be a social support resource. The theoretical framework of the nurse consolations will be based on Middle-range theory of self-care.

Outcome: Feasibility will be evaluated in terms of acceptability and adherence according to predefined feasibility criteria. The preliminary effect of the intervention on patient-reported outcomes, health behaviors and health outcomes will be evaluated in the intervention and the control group at baseline, one, three, six and twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for Ischemic heart disease (CABG or PCI), valve disease (TAVR, SAVR), and arrhythmia (ICD, pacemaker implantation or ablation) treated at Rigshospitalet and classified as high risk lonely according to the High Risk Loneliness (HiRL) tool

Exclusion Criteria:

* Patients who are unable to provide written consent, therefore, patients with severe cognitive or physical dysfunction will not be approached

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility, Acceptability | Measured at baseline
  Percentage of eligible patients who agree to participate in the trial
Feasibility, Adherence | 6 months follow-up after in-hospital cardiac treatment
  Percentage of patients in contact with the informal caregiver at least once a week face to face, by phone or virtually.

SECONDARY OUTCOMES:
Measure of social network members as informal caregivers | Measured at baseline
  Percentage of potential caregivers who accepts to be an informal caregiver
Measure of informal caregivers | 3 months follow-up after in-hospital cardiac treatment
  Percentage of informal caregivers participating in all three intervention consultations with the trial staff
Resource consumption | 6 months follow-up after in-hospital cardiac treatment
  Time resources used to complete the three nurse consultations

OTHER OUTCOMES:
Loneliness | Baseline, one, three, six and twelve months
  High Risk Loneliness tool. 2 item. Screeningscore 0 to 2, with a higher score indicating worse outcome
Self-care | Baseline, one, three, six and twelve months
  Self Care Self-Efficacy scale. 10 item scale answered on a Likert scale 1 to 5 with a lower score indicating worse outcome
Health-related quality of life | Baseline, one, three, six and twelve months
  HeartQoL. 10 item scale answered on a Likert scale 0-5, with a higher score indicating worse outcome
Anxiety and Depression | Baseline, one, three, six and twelve months
  Hospital Anxiety and Depression scale (HADS). 14 item scale. The scale offers two scores, HADS-A (anxiety) and HADS-D (depression). Answered in a Likert scale with a higher score indicating worse outcome
Health behaviors | Baseline, one, three, six and twelve months
  Smoking, alcohol consumption, weight, physical activity, participation in cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Selina K Berg, Professor, Principal Investigator — Rigshospitalet, Denmark; Mitti Blakø, PhD, Study Director — Rigshospitalet, Denmark; Anne V Christensen, PhD, Study Chair — Rigshospitalet, Denmark; Pernille Palm, PhD, Study Chair — Rigshospitalet, Denmark; Ida E Hojskov, PhD, Study Chair — Rigshospitalet, Denmark; Camilla Bernild, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Blakoe M, Olesen CS, Christensen AV, Palm P, Hoejskov IE, Berg SK. The rise and fall of a social support intervention feasibility trial targeting loneliness in patients with cardiac disease - lessons learned and future perspectives. BMC Nurs. 2024 Jun 24;23(1):423. doi: 10.1186/s12912-024-02113-6. PMID 38910234
- [Derived] Blako M, Christensen AV, Hojskov IE, Palm P, Berg SK. Protocol for a feasibility randomized trial of a social support intervention plus usual care versus usual care, targeting patients treated for cardiac disease who experience loneliness. Pilot Feasibility Stud. 2023 Feb 6;9(1):22. doi: 10.1186/s40814-023-01255-9. PMID 36747245